CLINICAL TRIAL: NCT03260153
Title: Deproteinised Calf Blood Serum Injection for the Treatment of Acute Intracerebral Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Stroke Association (Unknown)
Responsible Party: Principal Investigator, Xingquan Zhao, Professor of Neurology and Stroke Center, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBS-ICH
Record Dates: First submitted 2017-01-05; First posted 2017-08-24 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Perihematomal edema; Deproteinised Calf Blood Serum Injection
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deproteinised Calf Blood Serum Injection (Experimental): Participants will be randomly assigned to receive Deproteinised Calf Blood Serum Injection or placebo within 1 hour after randomization, once a day for 14 days.
  Interventions: Drug: Deproteinised Calf Blood Serum Injection
- Sodium Chloride Physiological Solution (Placebo Comparator): Participants will be randomly assigned to receive Deproteinised Calf Blood Serum Injection or placebo within 1 hour after randomization, once a day for 14 days.
  Interventions: Drug: Placebo (Sodium Chloride)

INTERVENTIONS:
Drug: Deproteinised Calf Blood Serum Injection
  Arms: Deproteinised Calf Blood Serum Injection
Drug: Placebo (Sodium Chloride)
  Arms: Sodium Chloride Physiological Solution

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of Deproteinised Calf Blood Serum Injection in alleviating perihematomal edema (PHE) and secondary brain injury, as well as neurologic deficits in patients with acute intracerebral hemorrhage (ICH).

DETAILED DESCRIPTION:
The study hypothesized that administration of Deproteinised Calf Blood Serum Injection would alleviate PHE and secondary brain injury, thus improving clinical outcomes in patients with ICH. The investigators will enroll 60 acute supratentorial ICH patients. Patients will be assigned randomly to receive either Deproteinised Calf Blood Serum Injection or placebo treatment, which is blinded to evaluator and patients. All patients in the study will receive standard care treatment and clinical, diagnostic, laboratory, safety, and follow-up evaluations. Blood will be drawn and brain MRI will be done in different time course. Follow-up evaluations, including National Institute of Health stroke scale(NIHSS), Stroke impact scale , Glasgow Coma Scale ,Barthel index score and modified Rankin scale assessments, will be done periodically until 90 days after onset.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of spontaneous intracerebral hemorrhage(sICH)
2. Bleeding into deep gray matter (basal ganglionic and thalamus), and the amount of bleeding between 5 and 30 ml;
3. Age between 18 and 80 years;
4. Presentation within 48 hours of symptom onset, and NCCT at 24 hours need to be done in patients presenting within 24 hours of symptom onset in order to exclude hematoma expansion.
5. Informed consent by patients or relatives.

Exclusion Criteria:

1. Â secondary ICH (secondary to trauma, tumor, vascular malformations, ischemic stroke hemorrhagic transformation, etc.);
2. Glasgow Coma Score of 3-8 at admission;
3. Parenchymal hemorrhage with ventricle involved;
4. Patients with hematoma expansion; .
5. Planned surgery within 3 days of symptom onset;
6. Incompletely absorbed brain hematoma previously;
7. Prestroke modified Rankin score(mRS)>1;
8. Patients with hemorrhagic disease or coagulation disorders;
9. Patients with severe liver and renal insufficiency;.
10. Patients with severe heart failure or other serious systemic diseases;
11. Patients with malignant tumors or ongoing anti-tumor therapy;
12. Patients with a history of dementia or mental disorders;
13. Pregnant or lactating women or those who has a recent fertility plan;
14. Any contraindications to MRI(such as cardiac pacemakers and other metal implants, claustrophobia);
15. Any other neuroprotective has been applied before randomization;
16. Terminal patients whose life expectancy <90 days;
17. Patients participating in other clinical trials 30 days prior to randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes of cytotoxic and vasogenic edema on day 3 and day 7-10 (MRI evaluation) | day 3, day 7-10
Changes of vasogenic edema on day 14 (CT evaluation) | day 14
Changes of the biomarkers（MMP3、MMP9、TNF-α、IL-6、CRP） in the peripheral blood on different time course. | at admission, day 3，day 3-7，day 14，day 30, day 90

SECONDARY OUTCOMES:
Clinical outcome evaluated by Glasgow Coma Scale(GCS)scores. | at admission, day 14， day 30， day 90
Clinical outcome evaluated by NIH Stroke Scale(NIHSS)scores. | at admission, day 14， day 30， day 90
Clinical outcome evaluated by Barthel Index(BI) scores. | day 14， day 30， day 90
Clinical outcome evaluated by Modified Rankin Scale(mRS)scores. | at admission, day 14， day 30， day 90
Clinical outcome evaluated by Stroke Impact Scale (SIS) scores. | day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality, China